CLINICAL TRIAL: NCT05143021
Title: Sickle Cell Disease Obstetric Multi-Disciplinary Care Programme: Prospective Multi-Centre Cohort Study
Brief Title: Sickle Cell Disease Obstetric Multi-Disciplinary Care Programme
Acronym: SCOB-II
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Michael DeBaun, Director of Vanderbilt-Meharry Center of Excellence for Sickle Cell Disease, Vanderbilt University Medical Center
Other Study IDs: 211778
Record Dates: First submitted 2021-11-19; First posted 2021-12-03 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease; Pregnancy Related
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant Women with Sickle Cell Disease: Pregnant women with sickle cell disease from the 3 centers in Ghana
  Interventions: Other: Multidisciplinary Sickle Cell Disease- Obstetric Team

INTERVENTIONS:
Other: Multidisciplinary Sickle Cell Disease- Obstetric Team — Modified multidisciplinary teams for pregnant women with sickle cell disease including members from an obstetrics team and sickle cell disease team.

SUMMARY:
To implement an effective but low-cost strategy to decrease SCD maternal and perinatal mortality in Ghana. The objectives are to 1) assess the impact of a multidisciplinary SCD-obstetric team for decreasing mortality across three hospital sites in Ghana. 2) assess the implementation fidelity for 2a) preventing and 2b) treating acute chest syndrome in pregnant women with SCD admitted to the hospital. 3) standardize an ultrasound protocol for the prospective monitoring of fetal growth among pregnant women with SCD.

DETAILED DESCRIPTION:
Ghana, has a high burden of sickle cell disease (SCD), with a disproportionately high maternal and perinatal morbidity and mortality. In 2015, the investigators established a multidisciplinary SCD Obstetrics team to implement low-technology evidence-based protocols (EBP) to prevent and treat acute chest syndrome (ACS), which is the leading cause of maternal death, institute maternal and fetal monitoring, and ensure better-coordinated care for in-patients. These interventions resulted in an 89.1% risk reduction in maternal mortality over 13 months. The investigators have designed an implementation protocol that allows for the systematic tailoring and implementation of this EBP at facilities that employ few (or no) specialized physicians.

The critical and unanswered question is: can the dramatic reduction in maternal and perinatal mortalities observed at KBTH be maintained and replicated with high fidelity at other tertiary hospitals in Ghana? This study, set in a region with the world's highest SCD prevalence, has the potential to impact maternal and neonatal mortality by tailoring evidence-based protocols to facilitate use by non-specialized health care providers. This project has the potential to change the way pregnant women with SCD are managed in Ghana and the rest of sub-Saharan Africa. If successful, this study will form a blueprint for the scale-up of this evidence-based protocol across the country and the West Africa sub-region, where pregnant women with SCD face an uncertain future. Additionally, the project can serve as a model for training clinical researchers, public health, and social scientists in implementation science for major interventions in maternal and perinatal health in Ghana.

The investigators propose a standards care prospective protocol to test the following two primary hypotheses:

1. After implementing a hospital-tailored task-shifting intervention program in the tertiary hospitals, there will be a 60% relative risk reduction in maternal mortality among pregnant women with SCD.
2. A. There will be at least a 90% fidelity to evidence-based guidelines for the prevention of ACS for women with SCD at high risk for ACS (acute pain and post-surgery) B. There will be at least a 90% fidelity to evidence-based guidelines for the treatment of ACS for women with SCD at high risk for ACS (acute pain and post-surgery)

This will be a multi-center prospective cohort study involving pregnant women with SCD who attend antenatal care at three referral hospitals. Participants will be enrolled from the booking visit over 18 months and managed with the evidence-based clinical guidelines plus multi-disciplinary team standard care protocol and followed up prospectively until delivery and up to six weeks after delivery.

ELIGIBILITY:
Inclusion Criteria:

* All study participants will be adults between the reproductive ages of 18 to 45 years as defined by World Health Organization (WHO)
* Confirmed SCD status by Hb-electrophoresis in alkaline medium
* Pregnancy should be confirmed by urine or blood pregnancy test and pelvic ultrasound scan.

Exclusion Criteria:

* All pregnant women without a confirmed Hb phenotype or electrophoresis report
* All pregnant women with SCD who present to the Greater Accra Regional Hospital or Tamale Teaching Hospital for acute admissions, labor, and delivery
* All pregnant women with SCD with undetermined Hb phenotypes on Hb electrophoresis.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women and their health care providers living with SCD in Ghana (Accra-Tema metropolis and Tamale).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Maternal and Perinatal Mortality Rates | Baseline- 6 weeks post delivery
  Change in maternal and perinatal mortality rates in the pre-implementation and post-implementation phases.
The Fidelity to the Evidence-Based Guidelines | Baseline- 6 weeks post delivery
  Fidelity to the evidence-based guidelines for the prevention of acute chest syndrome in pregnant women with SCD utilizing a questionnaire.
Participants with Acute Chest Syndrome | Baseline- 6 weeks post delivery
  The proportion of participants with ACS (based on diagnostic criteria) who are appropriately identified and treated.
The Fidelity to the Standardized Ultrasound Protocol | Baseline- 6 weeks post delivery
  The fidelity to the standardized ultrasound protocol for detection of Small for Gestational Age (SGA) or Intrauterine Growth Restriction (IUGR) in pregnant women with SCD utilizing a questionnaire.
Maternal Nutrition Supply Association to Fetus | Baseline- 6 weeks post delivery
  Affect of maternal nutrition supply on fetus (maternal diet, cataloged in a questionnaire) on birth weight and adverse birth outcomes.
Maternal Nutrition Supply Association to Fetus | Baseline- 6 weeks post delivery
  Affect of maternal nutrition supply on fetus (pre-pregnancy body mass index, measured in kilograms and height in meters) on birth weight and adverse birth outcomes.
Maternal Nutrition Supply Association to Fetus | Baseline- 6 weeks post delivery
  Affect of maternal nutrition supply on fetus (gestational weight gain, measured in kilograms) on birth weight and adverse birth outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Leshana St. Jean, PhD, Study Director — Vanderbilt University Medical Center
Locations (3):
- Ghana (3):
  - Greater Accra Regional Hospital, Accra
  - Korle Bu Teaching Hospital, Accra
  - Tamale Teaching Hospital, Tamale

IPD SHARING:
Plan to Share IPD: No